CLINICAL TRIAL: NCT04031456
Title: Investigating Reactivation of Ovarian Function Following Autologous PRP Intra-ovarian Infusion in POI Patients
Brief Title: Autologous PRP Infusion May Restore Ovarian Function and May Promote Folliculogenesis in POI Patients
Acronym: PRP
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genesis Athens Clinic (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRP- POI
Record Dates: First submitted 2017-10-25; First posted 2019-07-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Menopause, Premature; Menopause Related Conditions; Menopausal Syndrome; Premature Ovarian Failure; Ovarian Failure, Premature
MeSH Terms: conditions — Menopause, Premature; Primary Ovarian Insufficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving PRP treatment (Experimental): Women presenting with POI, 25-39 years of age, treated with autologous PRP intra ovarian infusion
  Interventions: Biological: Autologous Platelet Rich Plasma
- Participants receiving Platelet Free Plasma (PFP) treatment (Placebo Comparator): Women presenting with POI, 25-39 years of age, treated with autologous PFP intra ovarian infusion
  Interventions: Biological: Placebo-Platelet Free Plasma

INTERVENTIONS:
Biological: Autologous Platelet Rich Plasma — Autologous PRP intra ovarian infusion
  Other Names: PRP; Platelet Rich Plasma
  Arms: Participants receiving PRP treatment
Biological: Placebo-Platelet Free Plasma — Autologous PFP intra ovarian infusion
  Other Names: PFP
  Arms: Participants receiving Platelet Free Plasma (PFP) treatment

SUMMARY:
Autologous PRP intra ovarian infusion may restore ovarian function, may promote folliculogenesis and may improve patients' hormonal profile in patients presenting with POI.

DETAILED DESCRIPTION:
This triple-blind Randomized Controlled Trial (RCT) aims to investigate the effectiveness of autologous PRP intra ovarian infusion on reactivating ovarian functionality and on promoting folliculogenesis in regard to patients presenting with POI. PRP is blood plasma prepared from fresh whole blood that has been enriched with platelets. It is collected from peripheral veins and contains several growth factors such as vascular endothelial growth factor (VEGF), epidermal growth factor (EGF), platelet derived growth factor (PDGF), transforming growth factor (TGF) and other cytokines all of which stimulate tissue proliferation and growth. PRP has been employed in several medical conditions in Orthopedics, Dermatology, and Ophthalmology for wound healing. It's efficacy in ovarian rejuvenation and reactivation and endometrial regeneration has not been fully elucidated. This study aims to investigate the effect of autologous PRP intra ovarian infusion on restoring ovarian tissue functionality in POI patients.

ELIGIBILITY:
Inclusion Criteria:

* Age < 40 years, presenting with amenorrhea or menstrual cycle irregularities for at least four months, and elevated FSH levels >25 IU/L recorded on two occasions >4 weeks apart
* Normal Karyotype: 46, XX
* Discontinuation of any complementary/adjuvant treatment including hormone replacement, acupuncture, and botanotherapy, for at least three months prior to recruitment.
* Willing to comply with study requirements

Exclusion Criteria:

* Any pathological disorder related to reproductive system anatomy
* AMH > 8 pmol/L
* Endometriosis
* Adenomyosis
* Fibroids and adhesions
* Infections in reproductive system
* Current or previous diagnosis of cancer in reproductive system
* History of familiar cancer in reproductive system
* Severe male factor infertility
* Prior referral for PGT
* Ovarian inaccessibility
* Endocrinological disorders (Hypothalamus-Pituitary disorders, thyroid dysfunction, diabetes mellitus, metabolic syndrome)
* BMI>30 kg/m2 or BMI<18.5 kg/m2
* Systematic autoimmune disorders

Ages: 25 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Restoration of menstrual cycle | Three months
  Regular menstrual cycle
Serum FSH levels | Follow-up period of three months entailing monthly evaluation
  Serum FSH levels evaluated monthly for three consecutive months

SECONDARY OUTCOMES:
Serum AMH levels | Follow-up period of three months entailing monthly evaluation
  Serum ΑΜΗ levels evaluated monthly for three consecutive months
Serum LH levels | Follow-up period of three months entailing monthly evaluation
  Serum LH levels evaluated monthly for three consecutive months
Serum Estradiol levels | Follow-up period of three months entailing monthly evaluation
  Serum estradiol levels evaluated monthly for three consecutive months
Serum Progesteron levels | Follow-up period of three months entailing monthly evaluation
  Serum progesterone levels evaluated monthly for three consecutive months
Antral Follicle Count (AFC) | Follow-up period of three months entailing monthly evaluation
  AFC evaluated monthly, on day 2 of the menstrual cycle, for three consecutive months

CONTACTS AND LOCATIONS:
Locations (1):
- Genesis AC, Athens, Greece